CLINICAL TRIAL: NCT01953835
Title: A Two-part Healthy Volunteer Study to Investigate Both the Interaction of GSK2586184 With Rosuvastatin and Simvastatin and to Compare the Pharmacokinetics of Two Different Formulations of GSK2586184
Brief Title: A Two-part Study to Investigate the Interaction and Pharmacokinetics of GSK2586184
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 117171
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Pharmacokinetics; GSK2586184; Simvastatin; Rosuvastatin; Poloxamer
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Simvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Cohort A is a single-sequence, open-label study in which each subject will receive Simvastatin 10 mg single dose oral tablet on Days 1 and 10, Rosuvastatin 10 mg single dose oral tablet on Days 3 and 12 and GSK2586184 standard formulation 400 mg twice daily oral tablet from Day 6 to Day 14 immediately after food. At Day 10 GSK2586184 and Simvastatin and at Day 12, GSK2586184 and Rosuvastatin will be co-administered.
  Interventions: Drug: GSK2586184 standard formulation; Drug: Simvastatin; Drug: Rosuvastatin
- Cohort B (Experimental): Cohort B is a three-way crossover study in which each subject will receive a single dose of GSK2586184 standard formulation 400 mg oral tablet with food and two doses of a new formulation of GSK2586184 400 mg oral tablet, once with food and once in a fasted state, on Day 1, 4 and 7 according to their treatment sequence, with a 3-day wash out between doses.
  Interventions: Drug: GSK2586184 standard formulation; Drug: GSK2586184 new formulation

INTERVENTIONS:
Drug: GSK2586184 standard formulation — GSK2586184 standard formulation is a white film coated round biconvex 200 mg oral tablet. For cohort A, it is to be administered at 400 mg (200 mg x 2 tablets) twice daily from Day 6 to Day 14. For cohort B, it is to be administered at 400 mg (200 mg x 2 tablets) single dose after standard breakfast either on Day 1, 4 and 7 according to the treatment sequence, each separated by a 3-day wash out period.
Drug: Simvastatin — Simvastatin 10 mg oral tablet is peach-coloured, oval-shaped tablets. It is to be administered orally as a single dose of 10 mg tablet on the mornings of Day 1 and Day 10.
  Arms: Cohort A
Drug: Rosuvastatin — GSK2586184 new formulation without poloxamer is a white film coated round biconvex 200 mg oral tablet. In cohort B, it is to be administered at 400 mg (200 mg x 2 tablets) single dose once after standard breakfast and once after overnight fasting, either on Day 1, 4 and 7 according to the treatment sequence, each separated by a 3-day washout period.
  Arms: Cohort A
Drug: GSK2586184 new formulation — GSK2586184 new formulation without poloxamer is a white film coated round biconvex 200 mg oral tablet. In cohort B, it is to be administered at 400 mg (200 mg x 2 tablets) single dose once after standard breakfast and once after overnight fasting, either on Day 1, 4 and 7 according to the treatment sequence, each separated by a 3-day washout period.
  Arms: Cohort B

SUMMARY:
This study is a Phase I, two-part, open-label study designed to evaluate the effect of repeated doses of GSK2586184 on the pharmacokinetics (PK) of Simvastatin and Rosuvastatin in healthy volunteers (Cohort A), and to evaluate the pharmacokinetics of a new tablet formulation of GSK2586184 in healthy male volunteers (Cohort B). Cohort A is a single sequence drug interaction study in which 28 subjects (14 female and 14 male subjects) will be enrolled. Each subject will receive single doses of Simvastatin and Rosuvastatin on two occasions, once alone and once following administration of repeated doses of GSK2586184. Cohort B is a 3-way crossover PK study in which 9 male subjects will be randomized (3 subjects to each treatment sequence). Each subject will receive a single dose of the standard formulation of GSK2586184 with food and two doses of a new formulation of GSK2586184, once with food and once in a fasted state, according to their treatment sequence, with a 3-day wash out between doses. The primary aim of the study is to investigate the effects of GSK2586184 on the pharmacokinetics of the 2 statins and to assess the impact of dosing with and without food on a new formulation of GSK2586184 tablet.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent. (Females are only eligible for Cohort A).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with Hemoglobin (Hgb), Hematocrit (HCT), White blood cells (WBC), neutrophil or platelet values outside the normal range should always be excluded from enrolment.
* Body Mass Index (BMI) within the range 18 - 30 Kilogram per meter square (kg/m^2) (inclusive).
* For Cohort A only, a female subject is eligible to participate if she is of non-childbearing potential, defined as: Pre-menopausal females with a documented tubal ligation, tubal occlusion procedure followed by a hysterosalpingogram that confirmed bilateral tubal occlusion, bilateral salpingectomy or hysterectomy [ "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter mIU/mL and estradiol < 40 picogram/milliliter (pg/mL) (<147 picomole/liter is confirmatory].
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods: Condom plus partner use of a highly effective contraceptive or abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. This criterion must be followed from the time of the first dose of study medication and for at least 2 weeks after their last dose.
* Normal creatinine clearance values at screening (calculated from serum creatinine by a predicting equation using Cockcroft-Gault formula), normal serum creatinine value as defined by the local reference laboratory, normal urine microscopy and no significant proteinuria on dipstick testing.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <= 1.5 x Upper Limit of Normal [ULN] (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35 %).
* Based on averaged QT duration corrected for heart rate by Fridericia's formula (QTcF) values of triplicate ECGs obtained over a brief recording period: QTcF < 450 millisecond (msec); or QTcF < 480 msec in subjects with Bundle Branch Block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Criteria Based Upon Medical Histories

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects who have taken statins and/or other Organic Anion-Transporting Polypeptide (OATP) and Breast Cancer Resistance Protein (BCRP) sensitive substrates (e.g. rapaglinide) in the 4 weeks prior to screening.
* A live vaccination within 4 weeks before the first dose of study medication, or a live vaccination planned during the course of the study (until completion of the follow-up visit).
* For Cohort A only: Any subject who has received an allogeneic bone marrow transplant must be excluded.

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* Glycosylated Haemoglobin (HbA1c) result > 6.5 % (or 48 mmol/mol)
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10-04 (Actual); Primary Completion 2014-03-10 (Actual); Study Completion 2014-03-10 (Actual)

PRIMARY OUTCOMES:
Cohort A: AUC (zero to infinity), AUC (0-t) and Cmax of Rosuvastatin alone and in the presence of GSK2586184 | Days 3 and 12 (1 hour (h) pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours (hrs) post-dose)
  Blood samples will be collected to analyse PK parameters of Rosuvastatin including area under the plasma concentration-time curve from time zero to infinity [AUC(0-inf)], area under the plasma concentration-time curve from time zero to the last quantifiable concentration [AUC(0-t)] and the maximum observed plasma concentration (Cmax).
Cohort A: AUC (zero to infinity), AUC(0-t) and Cmax of Simvastatin/Simvastatin acid alone and in the presence of GSK2586184. | Days 1 and 10 (1 h pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24 and 48 hrs post-dose)
  Blood samples will be collected to analyse PK parameters of Simvastatin including AUC(0-inf), AUC(0-t) and Cmax.
Cohort B: AUC (zero to infinity), AUC(0-24), Tmax and Cmax of GSK2586184 (standard formulation, containing poloxamer) and GSK2586184 (new formulation, without-poloxamer). | Day 1, 4 (1 h pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hrs post dose) and Day 7 (1 h pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, and 24)
  Blood samples will be collected to analyse PK parameters of GSK2586184 (standard and new formulation) including AUC(0-inf), area under the plasma concentration-time curve from time 0 to 24 hrs (AUC(0-24)), time to maximum observed plasma drug concentration (Tmax) and Cmax.
Cohort B: AUC(zero to infinity), AUC(0-24), Tmax and Cmax of GSK2586184 (new formulation, without-poloxamer) dosed with and without food. | Day 1, 4 (1 h pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hrs post dose) and Day 7 (1 h pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, and 24)
  Blood samples will be collected to analyse PK parameters of GSK2586184 (new formulation, without-poloxamer) including AUC (0-inf), AUC(0-24), Tmax and Cmax.

SECONDARY OUTCOMES:
Cohort A: AUC(0-12) and Cmax of GSK2586184 at steady state | Day 9 (1 h pre-dose, and 0.5, 1, 2, 4, 6, 8, 10 and 12 hrs post dose)
  Blood samples will be collected to analyse PK parameters of GSK2586184 at steady state including area under the plasma concentration-time curve from time 0 to 12 h (AUC (0-12)) and Cmax.
Cohort A: AUC (0-12) and Cmax of two metabolites of GSK2586184 (GSK2983628 and GSK3100466) at steady state | Day 9 (1 h pre-dose, and 0.5, 1, 2, 4, 6, 8, 10 and 12 hrs post dose)
  Blood samples will be collected to analyse PK parameters of GSK2983628 and GSK3100466 at steady state including AUC (0-12) and Cmax.
Cohort B: AUC (zero to infinity), AUC(0-24), Cmax, Tmax and t1/2 of two metabolites of GSK2586184 (GSK2983628 and GSK3100466) | Day 1, 4 (1 h pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hrs post dose) and Day 7 (1 h pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, and 24)
  Blood samples will be collected to analyse PK parameters of GSK2983628 and GSK3100466 including AUC (0-inf), AUC (0-24), Cmax, Tmax and terminal phase half-life (t1/2).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20846

REFERENCES:
- See also: Results for study 117171 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117171?search=study&search_terms=117171#rs